CLINICAL TRIAL: NCT03776578
Title: Prospective Proactive Swallowing Rehabilitation and Swallow Outcome for Advanced Oral Cancer Patients Treated With Wide Excision and Free Flap Reconstruction
Brief Title: Oral Cancer With Wide Excision and Free Flap Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201807023RINA
Record Dates: First submitted 2018-12-04; First posted 2018-12-14 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Head and neck Cancer surgery not treatment and rehabilitation: The patients with oral cavity cancer who weren't treated by radical operation and free flap reconstruction,and can't provide them with preventive swallowing rehabilitation
- Head and neck Cancer surgery treatment and rehabilitation: Head and neck cancer treatment has developed over the last decade, with improved mortality and survival rates, It is well accepted that pre-treatment swallow function is indicative of post-treatment status and is helpful in identifying patients with high risk of aspiration and dysphagia.Preventive swallowing rehabilitation including evaluation patient's swallowing function and propose rehabilitation and adaptive maneuver or change in food texture. The aim is to ensure safe swallowing and prevent deglutitive muscles from deconditioning. Investigators include patients with advanced oral cavity cancer who were treated by radical operation and free flap reconstruction, and provided them with preventive swallowing rehabilitation.Investigators then analyze the swallowing function, oral intake status, and nasogastric tube dependence rate and tracheostomy tube dependence rate.
  Interventions: Procedure: swallow fuction and swallow training

INTERVENTIONS:
Procedure: swallow fuction and swallow training — nasogastric tube dependence rate
  Groups: Head and neck Cancer surgery treatment and rehabilitation

SUMMARY:
A proactive speech-language pathologist program can be successfully established as part of the multidisciplinary care of patients with head and neck squamous cell carcinoma and improve patient quality of life.

DETAILED DESCRIPTION:
Head and neck cancer treatment has developed over the last decade, with improved mortality and survival rates, but the treatments often result in dysphagia (a difficulty in swallowing) as a side effect. Swallowing function is affected by the tumor itself, surgical resection of the lesion and neoadjuvant chemoradiation therapy. It is well accepted that pre-treatment swallow function is indicative of post-treatment status and is helpful in identifying patients with high risk of aspiration and dysphagia. In recent years, the concept of "use it, or lose it" has been widely advocated by specialists. Preventive swallowing rehabilitation including evaluation patient's swallowing function and propose rehabilitation and adaptive maneuver or change in food texture. The aim is to ensure safe swallowing and prevent deglutitive muscles from deconditioning. Moreover, aspiration can be prevented and adequate nutrition was maintained through the cancer treatment course. Investigators include patients with advanced oral cavity cancer who were treated by radical operation and free flap reconstruction, and provided them with preventive swallowing rehabilitation. Investigators then analyze the swallowing function, oral intake status, and nasogastric tube dependence rate and tracheostomy tube dependence rate.The participants received interventions as part of our routine medical care, and Investigators studied the effect of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Advanced Oral Cancer Patients Treated with Wide Excision and Free Flap Reconstruction

Exclusion Criteria:

Not willing to participate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For all outcome measures, descriptive statistics were generated. Statistical analysis will be performed using the Statistical Package of Social Sciences (SPSS) software version 23.0.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
nasogastric tube dependence rate | 2 years
  nasogastric tube dependence rate

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Hsuan Tseng, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Wen-Hsuan Tseng, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
protocal,patient treantment course

REFERENCES:
- [Background] Goepfert RP, Lewin JS, Barrow MP, Gunn GB, Fuller CD, Beadle BM, Garden AS, Rosenthal DI, Kies MS, Papadimitrakopoulou V, Lai SY, Gross ND, Schwartz DL, Hutcheson KA. Long-Term, Prospective Performance of the MD Anderson Dysphagia Inventory in "Low-Intermediate Risk" Oropharyngeal Carcinoma After Intensity Modulated Radiation Therapy. Int J Radiat Oncol Biol Phys. 2017 Mar 15;97(4):700-708. doi: 10.1016/j.ijrobp.2016.06.010. Epub 2016 Jun 15. PMID 27485284
- [Background] Goepfert RP, Lewin JS, Barrow MP, Fuller CD, Lai SY, Song J, Hobbs BP, Gunn GB, Beadle BM, Rosenthal DI, Garden AS, Kies MS, Papadimitrakopoulou VA, Schwartz DL, Hutcheson KA. Predicting two-year longitudinal MD Anderson Dysphagia Inventory outcomes after intensity modulated radiotherapy for locoregionally advanced oropharyngeal carcinoma. Laryngoscope. 2017 Apr;127(4):842-848. doi: 10.1002/lary.26153. Epub 2016 Jul 21. PMID 27440393
- [Result] Perry A, Lee SH, Cotton S, Kennedy C. Therapeutic exercises for affecting post-treatment swallowing in people treated for advanced-stage head and neck cancers. Cochrane Database Syst Rev. 2016 Aug 26;2016(8):CD011112. doi: 10.1002/14651858.CD011112.pub2. PMID 27562477
- [Result] Kraaijenga SAC, Molen LV, Stuiver MM, Takes RP, Al-Mamgani A, Brekel MWMVD, Hilgers FJM. Efficacy of a novel swallowing exercise program for chronic dysphagia in long-term head and neck cancer survivors. Head Neck. 2017 Oct;39(10):1943-1961. doi: 10.1002/hed.24710. Epub 2017 Aug 2. PMID 28766850
- [Result] Ajmani GS, Nocon CC, Brockstein BE, Campbell NP, Kelly AB, Allison J, Bhayani MK. Association of a Proactive Swallowing Rehabilitation Program With Feeding Tube Placement in Patients Treated for Pharyngeal Cancer. JAMA Otolaryngol Head Neck Surg. 2018 Jun 1;144(6):483-488. doi: 10.1001/jamaoto.2018.0278. PMID 29710108